CLINICAL TRIAL: NCT07059832
Title: Application of 68Ga-NODAGA-SNA006 in Patients With Solid Tumor or Lymphoma
Brief Title: Application of 68Ga-NODAGA-SNA006 Positron Emission Tomography/Computed Tomography (PET/CT) in Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Yuxuan Zhao, Clinical Professor, First Hospital of China Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [2024]1161
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and safety of 68Ga-NODAGA-SNA006 (Experimental): 68Ga-NODAGA-SNA006 0.05 mCi/Kg, interval time between FDG was within five days
  Interventions: Drug: 68Ga-NODAGA-SNA006

INTERVENTIONS:
Drug: 68Ga-NODAGA-SNA006 — 68Ga-NODAGA-SNA006 PET/CT: after intravenous injection of 0.05 mCi/kg body weight of quality-controlled 68Ga-NODAGA-SNA006, an integrated PET/CT scanner (Biograph mCT; Siemens, Germany) will be applied.

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the safety and clinical predictive value of 68Ga-NODAGA-SNA006 in subjects with solid tumor or lymphoma.

DETAILED DESCRIPTION:
The aim of this study was to explore the safety and clinical predictive value of 68Ga-NODAGA-SNA006 in patients with solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who were diagnosed with malignant tumors;
2. Patients are between 18 and 80 years of age are between 18 and 80 years of age.

Exclusion Criteria:

1. Participants who were unable or unwilling to provide written informed consent.
2. Participants who were unable to successfully complete the examination and are forced to abort the test in the middle of the test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of 68Ga-NODAGA-SNA006-emergent Adverse Events | 3 YEAR
  Through PET/CT, Visual analysis was positive, or the SUVmax was more than the mediastinum
Biodistribution of 68Ga-NODAGA-SNA006 | 3 YEAR
  Through PET/CT analysis, SUVmax and SUVmean of the organs

SECONDARY OUTCOMES:
Correlation analysis of 68Ga-NODAGA-SNA006 uptake and tumor immune phenotype | 3 YEAR
  Correlation coefficients (r²) between SUVmax and SUVmean measured by PET/CT and immunophenotypes

CONTACTS AND LOCATIONS:
Overall Officials: li, Study Director — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China